CLINICAL TRIAL: NCT01092364
Title: Cell Phone Intervention in Young Adults
Acronym: CITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00024782; 1U01HL096720 (NIH)
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Obesity
Keywords: Young adults
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cell phone intervention (Experimental): Behavioral lifestyle intervention for weight loss, delivered by cell phone.
  Interventions: Behavioral: Behavioral weight loss intervention
- Personal counseling intervention (Experimental): Behavioral lifestyle intervention for weight loss, delivered by personal counseling.
  Interventions: Behavioral: Behavioral weight loss intervention
- Advice only (No Intervention): Advice only control group.

INTERVENTIONS:
Behavioral: Behavioral weight loss intervention — Behavioral lifestyle intervention for weight loss, compared to advice-only control.
  Arms: Cell phone intervention; Personal counseling intervention

SUMMARY:
Weight gain accelerates during early adulthood, and leads to the health consequences of obesity (high blood pressure, diabetes, heart disease, etc). Most weight loss studies enroll middle-aged adults. This study tests the hypothesis that a weight loss intervention that builds on prior research evidence but is enhanced with technological innovations will lead to weight loss in a diverse group of overweight and obese adults aged 18-35 years. The technology intervention, using cell phone applications, will be compared to an "advice only" control group and to a group receiving a more traditional personal coaching intervention.

DETAILED DESCRIPTION:
Trials in middle aged adults indicate that weight loss can be achieved and sustained with frequent contact over a long period of time, frequent self-monitoring, social support and motivational counseling. However, it is unclear whether this strategy would work in younger adults. Based on life stage, cultural context, environmental circumstances, and marketing pressures, behavioral intervention may need to be substantially modified to be effective in young adults. Even more adaptation will be required for intervention to be effective in young adults from racial/ethnic minority groups. The proposed intervention builds on prior evidence with innovations directed at increasing effectiveness in young adults.

Using cell phones to deliver a weight control intervention in this age group has the potential to be engaging, enjoyable, practical, cost-effective, sustainable, and broadly disseminated. We propose a trial in which a highly innovative but more risky intervention based almost entirely on use of cell phone technology and a second more incremental innovation over traditional behavioral intervention are each compared to a usual care control group. We will recruit a diverse target population of overweight/obese, generally healthy young adults, comprising approximately 35% non-Latino Whites, 35% non-Latino Blacks, and 30% Latinos, to be randomized to: 1) Usual care control: Educational materials and information but no behavioral intervention; 2) Cell-phone intervention: similar education and knowledge as the control group, but thereafter a behavioral intervention will be delivered almost exclusively via cell phone, particularly using the self-monitoring and social networking features of this technology; 3) Personal contact with cell-phone enhancement: personal contact intervention enhanced by cell-phone for self-monitoring.

The post-randomization intervention period will last 24 months. The primary outcome is change in weight 12 months post-randomization; an important secondary outcome is weight change at 24 months.

The formative phase will focus largely on technology/intervention development.

To assess maintenance of weight loss, after completion of the primary outcome assessment (24 months post-randomization), participants in the control group are followed observationally; those in the cell-phone and personal coaching interventions are re-randomized to either continue intervention or stop intervention with observational follow-up. All participants who agree to participate in this maintenance phase are followed for an additional 2-3 years with data collection every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years;
* BMI >=25;
* Using a cellphone.

Exclusion Criteria:

* Diabetes mellitus;
* Pregnant or nursing;
* Use of weight loss medications, systemic steroids, antipsychotics, or diabetes medication;
* Prior weight loss surgery;
* Cardiovascular (CVD) event in past 6 months;
* Current malignancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 365 (Actual)
Dates: Start 2010-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura P Svetkey, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Batch BC, Tyson C, Bagwell J, Corsino L, Intille S, Lin PH, Lazenka T, Bennett G, Bosworth HB, Voils C, Grambow S, Sutton A, Bordogna R, Pangborn M, Schwager J, Pilewski K, Caccia C, Burroughs J, Svetkey LP. Weight loss intervention for young adults using mobile technology: design and rationale of a randomized controlled trial - Cell Phone Intervention for You (CITY). Contemp Clin Trials. 2014 Mar;37(2):333-41. doi: 10.1016/j.cct.2014.01.003. Epub 2014 Jan 21. PMID 24462568
- [Background] Svetkey LP, Batch BC, Lin PH, Intille SS, Corsino L, Tyson CC, Bosworth HB, Grambow SC, Voils C, Loria C, Gallis JA, Schwager J, Bennett GG. Cell phone intervention for you (CITY): A randomized, controlled trial of behavioral weight loss intervention for young adults using mobile technology. Obesity (Silver Spring). 2015 Nov;23(11):2133-41. doi: 10.1002/oby.21226. PMID 26530929
- [Background] Lin PH, Intille S, Bennett G, Bosworth HB, Corsino L, Voils C, Grambow S, Lazenka T, Batch BC, Tyson C, Svetkey LP. Adaptive intervention design in mobile health: Intervention design and development in the Cell Phone Intervention for You trial. Clin Trials. 2015 Dec;12(6):634-45. doi: 10.1177/1740774515597222. Epub 2015 Jul 30. PMID 26229119
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Lin PH, Grambow S, Intille S, Gallis JA, Lazenka T, Bosworth H, Voils CL, Bennett GG, Batch B, Allen J, Corsino L, Tyson C, Svetkey L. The Association Between Engagement and Weight Loss Through Personal Coaching and Cell Phone Interventions in Young Adults: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Oct 18;6(10):e10471. doi: 10.2196/10471. PMID 30341051

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cell Phone Intervention | Personal Counseling Intervention | Advice Only
Started | 122 | 120 | 123
Completed | 104 | 104 | 105
Not Completed | 18 | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cell Phone Intervention | Personal Counseling Intervention | Advice Only | Total
Number analyzed (Participants) | 122 | 120 | 123 | 365
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 122 | 120 | 123 | 365
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (4.2) | 29.4 (4.3) | 29.6 (4.3) | 29.4 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 85 | 85 | 254
  Male | 38 | 35 | 38 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 5 | 21
  Not Hispanic or Latino | 113 | 113 | 118 | 344
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 5 | 2 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 42 | 48 | 42 | 132
  White | 68 | 65 | 70 | 203
  More than one race | 0 | 3 | 3 | 6
  Unknown or Not Reported | 6 | 1 | 3 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 122 | 120 | 123 | 365
Weight [Mean (Standard Deviation); unit: kg] | 102.4 (25.2) | 99.3 (23.4) | 101.3 (22.6) | 101.0 (23.7)
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 35.7 (8.2) | 34.9 (7.5) | 35.1 (7.5) | 35.2 (7.8)
Waist Circumference [Mean (Standard Deviation); unit: cm] — Population: Waist circumference is presented by gender.
  cm
    Males: number analyzed (Participants) | 38 | 35 | 38 | 111
    Males | 113.8 (17.9) | 111.5 (16.4) | 109.8 (14.6) | 111.7 (16.3)
    Females: number analyzed (Participants) | 84 | 85 | 85 | 254
    Females | 109.3 (18.4) | 107.4 (16.4) | 107.9 (15.7) | 108.2 (16.8)
Dietary intake [Mean (Standard Deviation); unit: Scores on the HEI scale] — The Healthy Eating Index (HEI) will be used to measure dietary intake. HEI assesses conformance to the Dietary Guidelines for Americans. HEI scores can range from 0 to 100, with 0 representing the least overall healthy diet, and 100 representing the most overall healthy diet.
  Scores on the HEI scale | 51.6 (4.2) | 50.8 (3.6) | 50.7 (4.4) | 51.0 (4.1)
Physical activity [Mean (Standard Deviation); unit: kcal/week] | 756.0 (846.1) | 1009.3 (1346.4) | 865.9 (1133.9) | 879.7 (1134.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Time Frame: Baseline and 24 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Cell Phone Intervention | Personal Counseling Intervention | Advice Only
Number analyzed (Participants) | 122 | 120 | 123
kg | -0.99 (6.2) | -2.6 (6.0) | -1.7 (8.3)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Cell Phone Intervention | Personal Counseling Intervention | Advice Only
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/120 | 0/123
Serious Adverse Events (participants affected / at risk) | 4/122 | 4/120 | 5/123
Other Adverse Events (participants affected / at risk) | 8/122 | 4/120 | 1/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cell Phone Intervention (N=122) | Personal Counseling Intervention (N=120) | Advice Only (N=123)
Cholecystectomy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Obstetric hospitalization (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2)
Other (General disorders) | 4 (4) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cell Phone Intervention (N=122) | Personal Counseling Intervention (N=120) | Advice Only (N=123)
Musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No